CLINICAL TRIAL: NCT00771966
Title: Radical Prostatectomy and Perioperative Fluid Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Morten Bundgaard-Nielsen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RCT_PROST_ORTO
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: patients with cancer in the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Standard treatment (Placebo Comparator)
  Interventions: Procedure: Standard therapy
- SV maximization (Active Comparator)
  Interventions: Procedure: Maximization of cardiac stroke volume with fluid infusion

INTERVENTIONS:
Procedure: Standard therapy — Standard therapy
  Arms: Standard treatment
Procedure: Maximization of cardiac stroke volume with fluid infusion — Maximization of cardiac stroke volume with fluid infusion
  Arms: SV maximization

SUMMARY:
The optimal amount of fluid a patient need under surgery is not clear. Both to much and to little fluid can damage the organ functions.

A strategy called "Goal directed therapy", where the fluid amount a patient need is guided by the stroke volume, has shown to minimize post-operative nausea and vomiting.

The investigators intend to investigate if patients treated after these standards, has a better outcome then patients treated after normal regimes, regarding post-operative orthostatic-intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer in there prostate

Exclusion Criteria:

* Patients who don't understand the information
* ASA > III
* Patients that are under treatment with the drug triazolam
* Patients with af known renal decease
* Patients with a psychiatric decease
* Alcohol abuse
* Severe haemorrhagic decease
* Cancer in the mouth,pharynx, larynx or oesophagus

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To investigate orthostatic cardiovascular response and orthostatic intolerance in patients after removal of the prostate | 6 hours

SECONDARY OUTCOMES:
Investigate intraoperative haemodynamics | Intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of anesthesiology, Rigshospitalet, Copenhagen, Denmark